CLINICAL TRIAL: NCT00540423
Title: Clinical Evaluation of SB-497115-GR in Chronic Idiopathic Thrombocytopenic Purpura (ITP) -A Multicenter Study in Subjects With Chronic ITP Receiving a Double-Blind, Placebo-Controlled, Short-Term Treatment Followed by an Open-Label, Uncontrolled, Long-Term Treatment- <Phase II/III Study>
Brief Title: Clinical Evaluation of SB-497115-GR in Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 108109
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Idiopathic Thrombocytopenic Purpura; Purpura, Thrombocytopenic, Idiopathic
Keywords: thrombopoietin,; immunosuppressive therapy,; eltrombopag,; idiopathic thrombocytopenic purpura,; blood platelet,; splenectomy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB-497115-GR group (Experimental): Subject will initiate treatment with SB-497115-GR 12.5mg once a day. Based on the subjects platelet count at each visit, the dose of SB-497115-GR may be adjusted at 12.5mg, 25mg or 50mg.
  Interventions: Drug: SB-497115-GR 12.5mg; Drug: SB-497115-GR 25mg; Drug: SB-497115-GR 50 mg
- placebo group (Placebo Comparator): Subject will initiate treatment with SB-497115-GR 12.5mg matching placebo once a day. Based on the subjects platelet count at each visit, the dose of SB-497115-GR 12.5mg matching placebo may be increased to 2 tablet of SB-497115-GR 12.5mg matching placebo.
  Interventions: Drug: SB-497115-GR 12.5mg matching placebo

INTERVENTIONS:
Drug: SB-497115-GR 12.5mg — SB-497115-GR 12.5mg tablet once a day
  Arms: SB-497115-GR group
Drug: SB-497115-GR 25mg — SB-497115-GR 25mg tablet once a day
  Arms: SB-497115-GR group
Drug: SB-497115-GR 12.5mg matching placebo — SB-497115-GR 12.5mg matching placebo x1 or 2 tablet once a day
  Arms: placebo group
Drug: SB-497115-GR 50 mg — SB-497115-GR 25mg tablet x2 once a day
  Other Names: SB-497115-GR 50mg
  Arms: SB-497115-GR group

SUMMARY:
This is a Phase II/III multicenter study comprising of the double-blind, followed by open-label phases to evaluate and compare the efficacy and tolerability of eltrombopag (SB-497115-GR) in chronic ITP patients

ELIGIBILITY:
Inclusion criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria.

At Screening (Week -4 or -3)

* Diagnosed with ITP for at least 6 months prior to screening.
* Have a platelet count of <30,000/µL.
* Previously treated refractory or relapsed patients who have failed to achieve a platelet count of >=30,000/µL despite one or more prior therapies (either H. pylori eradication, corticosteroids, splenectomy, danazol or immunosuppressive drugs). (Note: Previous H. pylori eradication must have been completed at least 3 months prior to screening and clearly be ineffective).
* Previous treatment for ITP with splenectomy, rituximab, and cyclophosphamide must have been completed at Week -4 and clearly be ineffective.
* Subjects treated with cyclosporine A, mycophenolate mofetil or danazol must be receiving a dose that has been stable for at least 3 months prior to screening."
* A complete blood count (CBC) within the reference range, with the following exceptions

  1. Hemoglobin: females >=9g/dL and males >=10g/dL are eligible for inclusion if hemorrhage is present.
  2. Neutrophil count >=1,500/µL (1.5x109/L) is required for inclusion.
* The following clinical chemistries MUST NOT exceed 1.2 times the normal reference range:creatinine, ALT, AST, total bilirubin and alkaline phosphatase.
* Albumin must be within 80 to 120% of normal range.
* Subject is >=20 years old.
* Female subjects must either be:
* of non-childbearing potential (bilateral tubal ligation or post-menopausal), or
* of childbearing potential and have a negative pregnancy test and agree to use contraceptive methods specified in the GSK List of Highly Effective Methods for Avoidance of Pregnancy
* Hospitalization status: No restriction.
* Gender: No restriction.
* Subject has signed and dated written informed consent. At Randomization (Week 0)
* Have a platelet count of <30,000/µL.
* Previous therapy for ITP with immunoglobulins (IVIG and anti-D) and vincristine must have been completed at least 2 weeks prior to randomization and the platelet count must show a clear downward trend after the last treatment with immunoglobulins.
* Subjects treated with corticosteroids or azathioprine must be receiving a dose that has been stable for at least 4 weeks prior to randomization.
* Prolongation of prothrombin time and activated partial thromboplastin time (aPTT) must not exceed 1.2 times the upper limit of the normal range with no history of hypercoagulable state. (Note: These parameters will be measured at screening or at randomization.)
* CBC and clinical chemistries fulfill the same criteria as those at screening.
* Reticulocyte count within the reference range or elevated in case of bleeding. (Note: This parameter will be measured at screening or at randomization.)

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study.

At Screening (Week -4 or -3)

* Any severe medical condition (cardiac, hepatic or renal disorder) other than chronic ITP. (Note: ""Severe"" is defined as >=Grade 3 as a rule according to the ""Classification of the Severity of Adverse Experiences (PAB/SD Notification No.80, dated 29 June 1992) (Appendix X).)
* History of suspected or confirmed arterial or venous thrombosis (e.g., myocardial infarction, deep vein thrombosis) within the last 1 year.
* History of drug/alcohol abuse or dependence within 1 year prior to screening.
* Previous treatment with SB-497115-GR.
* Suspected blood disorder other than ITP.
* Suspected platelet aggregation abnormality.
* Suspected cyclic thrombocytopenia
* Current or history of HIV infection or hepatitis B virus or hepatitis C virus infections.
* Current or history of malignancy (Exception: Subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible).
* Female subjects who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
* Subjects who are deemed unsuitable for the study by the investigator (or sub investigator).
* Subjects who are participating in any other clinical trials at present or ones who previously participated in clinical trials and were treated with investigational products within last one month." At Randomization (Week 0)
* Subject wishes to withdraw consent.
* Subject is lost to follow-up.
* Subject has consumed anti-platelet agents (e.g., ticlopidine and aspirin), anticoagulants, or non-steroidal anti-inflammatory drugs (NSAIDs) for 7days prior to the first dose of study medication and will require these medications during the study period.
* Subjects who are deemed unsuitable for the study by the investigator (or sub investigator).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Japan (6):
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Tomiyama Y, Miyakawa Y, Okamoto S, Katsutani S, Kimura A, Okoshi Y, Ninomiya H, Kosugi H, Nomura S, Ozaki K, Ikeda Y, Hattori T, Katsura K, Kanakura Y. A lower starting dose of eltrombopag is efficacious in Japanese patients with previously treated chronic immune thrombocytopenia. J Thromb Haemost. 2012 May;10(5):799-806. doi: 10.1111/j.1538-7836.2012.04695.x. PMID 22409309

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo 12.5 milligrams (mg) for the first 3 weeks of the double-blind phase. The dose of placebo was adjusted to 25 mg or 12.5 mg/day at Week 3 based on the participant's platelet count and then continued up to Week 7
- SB-497115-GR, Double-blind: SB-497115-GR 12.5 mg for the first 3 weeks of the double-blind phase. The dose of study medication was adjusted to 25 mg or 12.5 mg/day at Week 3 based on the participant's platelet count and then continued up to Week 7.
- SB-497115-GR, Open-label: All participants who received placebo and SB-497115-GR in the double-blind phase and completed the phase continued to receive SB-497115-GR in the open-label phase (19 weeks for SB-497115-GR group and 26 weeks for placebo group; all participants received 26 weeks in total). Dose adjustment to 12.5, 25, or 50 mg/day was allowed based on the participant's platelet count.
Period: Double-Blind Treatment Period
Arm/Group | Placebo | SB-497115-GR, Double-blind | SB-497115-GR, Open-label
Started | 8 | 15 | 0
Completed | 8 | 14 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Open-Label Treatment Period
Arm/Group | Placebo | SB-497115-GR, Double-blind | SB-497115-GR, Open-label
Started | 0 | 0 | 22
Completed | 0 | 0 | 20
Not Completed | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- SB-497115-GR: SB-497115-GR 12.5 mg for the first 3 weeks of the double-blind phase. The dose of study medication was adjusted at Week 3 based on the participant's platelet count and then continued up to Week 7.
- Placebo: Placebo 12.5 mg for the first 3 weeks of the double-blind phase. The dose of placebo was adjusted at Week 3 based on the participant's platelet count and then continued up to Week 7.
- Total: Total of all reporting groups
Arm/Group | SB-497115-GR | Placebo | Total
Number analyzed (Participants) | 15 | 8 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (13.72) | 58.4 (11.72) | 55.3 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 7 | 1 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese Heritage | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders at Week 6
Description: A responder was defined as a participant with a platelet count within the target range (>=50 x 10^9/Liter and <=400 x 10^9/Liter).
Time Frame: Week 6
Population: Full Analysis Set: all randomized participants, with the exception of (1) those who did not receive any dose of study medication and (2) those with no valid platelet count measurements on therapy
Measure: Number; unit: Participants
Arm/Group | SB-497115-GR | Placebo
Number analyzed (Participants) | 15 | 8
Participants
  Responders | 9 | 0
  Non-responders | 6 | 8
Statistical Analysis 1: Comparison: SB-497115-GR vs Placebo; Test type: Superiority or Other; Risk Difference (RD) = 60, 95% CI [35.21 to 84.79] — The units of risk difference is percentage

2. Secondary Outcome: Number of Participants Assessed as Responders in at Least 4 Assessments Between Weeks 2 and 6
Description: A responder was defined as a participant with a platelet count within the target range (>=50 x 10^9/Liter and <=400 x 10^9/Liter) at at least 4 out of 5 scheduled visits.
Time Frame: Weeks 2 through 6
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | SB-497115-GR | Placebo
Number analyzed (Participants) | 15 | 8
Participants
  Responders | 5 | 0
  Non-responders | 9 | 8

3. Primary Outcome: Percentage of Participants for Whom at Least 75% of Their Assessments During the Course of 26 Weeks of SB-497115-GR Treatment Met the Definition of Responders
Description: A responder was defined as a participant with a platelet count within the target range (>=50 x 10^9/Liter and <=400 x 10^9/Liter). Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Week 26
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- SB-497115-GR: SB-497115-GR during both the double-blind and open-label treatment phases
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
percentage of participants | 43.5
Statistical Analysis 1: Comparison: SB-497115-GR; Test type: Superiority or Other; Percentage of 75% responders = 43.5, 95% CI [23.19 to 65.51] — Confidence interval of the percentage of participants for whom at least 75% of their assessments during the course of 26 weeks of SB-494115-GR treatment met the definition of responders

4. Secondary Outcome: Percentage of Responders at Each Visit
Description: as for outcome 1
Time Frame: Days 8, 15, 22, 29, 36, and 43
Population: Full Analysis Set
Measure: Number; unit: Percentage of responders
Arm/Group | SB-497115-GR | Placebo
Number analyzed (Participants) | 15 | 8
Percentage of responders
  Day 8 | 6.7 | 0
  Day 15 | 26.7 | 0
  Day 22 | 33.3 | 0
  Day 29 | 60.0 | 0
  Day 36 | 66.7 | 0
  Day 43 | 60.0 | 0

5. Secondary Outcome: Mean Platelet Count at Each Visit
Description: Blood taken from peripheral blood vessels was used for the measurement of platelet counts.
Time Frame: Baseline and Days 8, 15, 22, 29, 36, and 43
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | SB-497115-GR | Placebo
Number analyzed (Participants) | 15 | 8
10^9/Liter
  Baseline | 19.3 (6.79) | 12.6 (8.65)
  Day 8 | 26.9 (17.77) | 14.3 (12.26)
  Day 15 | 54.9 (55.84) | 13.5 (12.15)
  Day 22 | 54.4 (46.88) | 11.6 (9.50)
  Day 29 | 73.3 (46.72) | 10.6 (9.04)
  Day 36 | 99.4 (78.62) | 11.9 (10.79)
  Day 43 | 95.1 (100.25) | 9.9 (4.76)

6. Secondary Outcome: Mean Change From Baseline in Platelet Counts at Each Visit
Description: Change from baseline was calculated as values at Days 8, 15, 22, 29, 36, and 43 minus baseline value
Time Frame: Baseline and Days 8, 15, 22, 29, 36, and 43
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Groups:
- SG-497115-GR: SB-497115-GR 12.5 mg for the first 3 weeks of the double-blind phase. The dose of study medication was adjusted at Week 3 based on the participant's platelet count and then continued up to Week 7.
Arm/Group | Placebo | SG-497115-GR
Number analyzed (Participants) | 8 | 15
10^9/Liter
  Day 8 | 1.6 (6.05) | 7.6 (16.47)
  Day 15 | 0.9 (5.46) | 35.5 (56.11)
  Day 22 | -1.0 (3.02) | 35.0 (46.52)
  Day 29 | -2.0 (4.17) | 53.9 (46.02)
  Day 36 | -0.8 (7.94) | 80.1 (77.06)
  Day 43 | -2.8 (9.41) | 75.8 (99.93)

7. Secondary Outcome: Percentage of Participants With Bleeding Episodes Since the Last Visit
Description: When abnormal bleeding(s) was found since the last visit, it was recorded as a bleeding episode(s).
Time Frame: Days 1, 8, 15, 22, 29, 36, and 43
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SB-497115-GR | Placebo
Number analyzed (Participants) | 15 | 8
Percentage of participants
  Day 1 | 33 | 75
  Day 8 | 13 | 63
  Day 15 | 14 | 63
  Day 22 | 29 | 75
  Day 29 | 0 | 38
  Day 36 | 7 | 63
  Day 43 | 14 | 75

8. Secondary Outcome: Number of Participants at Baseline and Days 8, 15, 22, 29, 36, and 43 of Treatment by Platelet Count Category
Description: Blood taken from peripheral blood vessels was used for the measurement of platelet counts.
Time Frame: Baseline and Days 8, 15, 22, 29, 36, and 43
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | SB-497115-GR | Placebo
Number analyzed (Participants) | 15 | 8
Participants
  Baseline, Platelet counts (PC) <=15 x 10^9/L | 3 | 6
  Baseline, PC >15 to <30 x 10^9/L | 12 | 2
  Baseline, PC >=30 to <=50 x 10^9/L | 0 | 0
  Baseline, PC =>50 to <=200 x 10^9/L | 0 | 0
  Baseline, PC >200 to <=400 x 10^9/L | 0 | 0
  Baseline, PC >400 x 10^9/L | 0 | 0
  Day 8, PC <=15 x 10^9/L | 3 | 5
  Day 8, PC >15 to <30 x 10^9/L | 6 | 2
  Day 8, PC >=30 to <=50 x 10^9/L | 5 | 1
  Day 8, PC =>50 to <=200 x 10^9/L | 1 | 0
  Day 8, PC >200 to <=400 x 10^9/L | 0 | 0
  Day 8, PC >400 x 10^9/L | 0 | 0
  Day 15, PC <=15 x 10^9/L | 2 | 6
  Day 15, PC >15 to <30 x 10^9/L | 3 | 1
  Day 15, PC >=30 to <=50 x 10^9/L | 5 | 1
  Day 15, PC =>50 to <=200 x 10^9/L | 3 | 0
  Day 15, PC >200 to <=400 x 10^9/L | 1 | 0
  Day 15, PC >400 x 10^9/L | 0 | 0
  Day 22, PC <=15 x 10^9/L | 3 | 5
  Day 22, PC >15 to <30 x 10^9/L | 3 | 3
  Day 22, PC >=30 to <=50 x 10^9/L | 3 | 0
  Day 22, PC =>50 to <=200 x 10^9/L | 5 | 0
  Day 22, PC >200 to <=400 x 10^9/L | 0 | 0
  Day 22, PC >400 x 10^9/L | 0 | 0
  Day 29, PC <=15 x 10^9/L | 1 | 6
  Day 29, PC >15 to <30 x 10^9/L | 0 | 2
  Day 29, PC >=30 to <=50 x 10^9/L | 4 | 0
  Day 29, PC =>50 to <=200 x 10^9/L | 9 | 0
  Day 29, PC >200 to <=400 x 10^9/L | 0 | 0
  Day 29, PC >400 x 10^9/L | 0 | 0
  Day 36, PC <=15 x 10^9/L | 2 | 7
  Day 36, PC >15 to <30 x 10^9/L | 0 | 0
  Day 36, PC >=30 to <=50 x 10^9/L | 2 | 1
  Day 36, PC =>50 to <=200 x 10^9/L | 9 | 0
  Day 36, PC >200 to <=400 x 10^9/L | 1 | 0
  Day 36, PC >400 x 10^9/L | 0 | 0
  Day 43, PC <=15 x 10^9/L | 2 | 7
  Day 43, PC >15 to <30 x 10^9/L | 2 | 1
  Day 43, PC >=30 to <=50 x 10^9/L | 1 | 0
  Day 43, PC =>50 to <=200 x 10^9/L | 7 | 0
  Day 43, PC >200 to <=400 x 10^9/L | 2 | 0
  Day 43, PC >400 x 10^9/L | 0 | 0

9. Secondary Outcome: Percentage of Responders at Each Visit
Description: as for outcome 3
Time Frame: Days 8, 15, 22, 29, 36, and 43; Weeks 10, 14, 18, 22, and 26
Population: Full Analysis Set
Measure: Number; unit: Percentage of responders
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
Percentage of responders
  Day 8 | 4.3
  Day 15 | 17.4
  Day 22 | 21.7
  Day 29 | 47.8
  Day 36 | 56.5
  Day 43 | 52.2
  Week 10 | 57.1
  Week 14 | 60.9
  Week 18 | 50.0
  Week 22 | 52.4
  Week 26 | 69.6

10. Secondary Outcome: Mean Platelet Counts of Participants at Each Visit
Description: Blood taken from peripheral blood vessels was used for the measurement of platelet counts. Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Baseline; Days 8, 15, 22, 29, 36, and 43; Weeks 10, 14, 18, 22, and 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
10^9/Liter
  Baseline | 16.5 (8.45)
  Day 8 | 23.0 (16.77)
  Day 15 | 41.5 (48.32)
  Day 22 | 41.0 (41.80)
  Day 29 | 55.3 (45.75)
  Day 36 | 78.1 (72.76)
  Day 43 | 78.0 (88.31)
  Week 10 | 88.9 (81.15)
  Week 14 | 121.6 (121.20)
  Week 18 | 87.3 (80.09)
  Week 22 | 78.5 (57.58)
  Week 26 | 86.2 (49.62)

11. Secondary Outcome: Mean Change From Baseline in Platelet Counts at Each Visit
Description: Change from baseline was calculated as values at Days 8, 15, 22, 29, 36, and 43 and Weeks 10, 14, 18, 22, and 26 minus baseline value. Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Baseline; Days 8, 15, 22, 29, 36, and 43; Weeks 10, 14, 18, 22, and 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
10^9/Liter
  Day 8 | 6.4 (13.53)
  Day 15 | 25.1 (46.73)
  Day 22 | 24.6 (39.37)
  Day 29 | 38.9 (42.37)
  Day 36 | 61.7 (69.53)
  Day 43 | 61.6 (86.72)
  Week 10 | 71.4 (80.01)
  Week 14 | 104.5 (120.20)
  Week 18 | 69.4 (80.23)
  Week 22 | 61.1 (54.85)
  Week 26 | 68.4 (46.49)

12. Secondary Outcome: Mean Maximum Duration for Which Participants Maintained Platelet Counts >=50 x 10^9/Liter and <=400 x 10^9/Liter
Description: Maximum duration is measured as the longest period (days) for which a participant continuously maintained platelet counts within the target range (>=50 x 10^9/Liter and <=400 x 10^9/Liter). Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Weeks 1 through 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
Days | 59.5 (46.99)

13. Secondary Outcome: Mean Total Time for Which Participants Maintained Platelet Counts >=50 x 10^9/Liter and <=400 x 10^9/Liter
Description: Total time is measured as the cumulative number of days over which platelet counts were maintained within the target range (>=50 x 10^9/Liter and <=400 x 10^9/Liter). Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Weeks 1 through 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
Days | 78.4 (54.56)

14. Secondary Outcome: Percentage of Participants With Bleeding Episode Since the Last Visit
Description: When abnormal bleeding(s) was found since the last visit, it was recorded as a bleeding episode(s). Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Days 1, 8, 15, 22, 29, 36, and 43; Weeks 10, 14, 18, 22, and 26
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
Percentage of participants
  Day 1 | 48
  Day 8 | 35
  Day 15 | 27
  Day 22 | 36
  Day 29 | 18
  Day 36 | 23
  Day 43 | 27
  Week 10 | 11
  Week 14 | 14
  Week 18 | 26
  Week 22 | 28
  Week 26 | 5

15. Secondary Outcome: Percentage of Participants With a Reduction in Dose and/or Number of Drugs of Concomitant ITP Medications From Baseline
Description: ITP medications are drugs, such as steroids or immunoglobulin, to be used for ITP. Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Baseline through Week 26
Population: Full Analysis Set. Four participants in the Full Analysis Set did not have concomitant ITP medication at Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 19
Percentage of participants | 36.8

16. Secondary Outcome: Percentage of Participants Who Received Rescue Treatment for ITP
Description: Rescue treatment for ITP is treatment applied to participants at high bleeding risk, such as those undergoing platelet transfusion or dose increase of steroids. Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Weeks 1 through 26
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
Percentage of participants | 9

17. Secondary Outcome: Mean Number of Days of Concomitant ITP Medication Use Per Month
Description: Cumulative number of days for which a participant received ITP medication during the treatment/total treatment period (months). Participants receiving placebo in the double-blind phase received SB-497115-GR in the open-label phase for up to 26 weeks. Participants receiving SB-497115-GR in the double-blind phase for 7 weeks continued to receive SB-497115-GR in the open-label phase for 19 weeks. The data from these two groups were pooled as a 26 week treatment of SB-497115-GR group and analyzed for the efficacy and safety.
Time Frame: Weeks 1 through 26
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SB-497115-GR
Number analyzed (Participants) | 23
Days | 25.14 (11.796)

18. Secondary Outcome: Pharmacokinetics of SB-497115-GR, Cmax
Description: Cmax: Peak plasma concentration of SB-497115
Time Frame: Week 9 or 10
Population: Pharmacokinetic (PK) Population: all participants with valid PK data following SB-497115-GR treatment
Measure: Mean (Standard Deviation); unit: ng/mL (nanograms/milliliter)
Groups:
- SB-497115-GR 12.5 mg: Participants who received 12.5 mg of SB-497115-GR on the PK sampling day
- SB-497115-GR 25 mg: Participants who received 25 mg of SB-497115-GR on the PK sampling day
- SB-497115-GR 50 mg: Participants who received 50 mg of SB-497115-GR on the PK sampling day
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 8 | 5 | 4
ng/mL (nanograms/milliliter) | 2992.4 (1253.14) | 6776.4 (2619.62) | 11877.8 (3926.21)

19. Secondary Outcome: Pharmacokinetics of SB-497115-GR, Tmax
Description: tmax: Time when Cmax was achieved
Time Frame: Week 9 or 10
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 8 | 5 | 4
Hours | 3.192 [2.00 to 4.17] | 4.000 [2.00 to 4.00] | 2.967 [1.92 to 4.17]

20. Secondary Outcome: Pharmacokinetics of SB-497115, t1/2
Description: t1/2 is half life based on the terminal phase
Time Frame: Week 9 or 10
Population: PK Population. Data from one participant were abnormal; this participant was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 7 | 5 | 4
Hours | 19.50 (7.164) | 29.96 (7.664) | 18.19 (4.938)

21. Secondary Outcome: Pharmacokinetics of SB-497115-GR, Lambda z
Description: Lambda z is first order rate constant associated with the terminal portion of the plasma concentration curve.
Time Frame: Week 9 or 10
Population: PK Population. Data from one participant were abnormal; this participant was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: 1/hour
Groups:
- SB-497115-GR 25 mg: Participants who received 25 mg of SB-497511-GR on the PK sampling day
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 7 | 5 | 4
1/hour | 0.04021 (0.015558) | 0.02724 (0.006881) | 0.04040 (0.011422)

22. Secondary Outcome: Pharmacokinetics of SB-497115-GR, AUClast and AUC0-24
Description: AUC is area under a concentration vs. time curve.
  AUC0-24 (Area under the plasma concentration-time curve between 0 to 24 hrs) is calculated using the following equation:
  AUC0-24= AUClast + Clast × (1 - e-λz × [24-tlast])/λz. AUClast is AUC (area under a curve) computed to the last observation. Clast is concentration of last observation.
Time Frame: Week 9 or 10
Population: PK Population. Data from one participant were abnormal; this participant was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- SB-497115-GR 12.5 mg: Participants who received 12.5 mg of SB-497511-GR on the PK sampling day
- SB-497115-GR 50 mg: Participants who received 50 mg of SB-497511-GR on the PK sampling day
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 7 | 5 | 4
hr*ng/mL
  AUClast | 41671.5 (24344.64) | 92556.2 (41095.63) | 171523.2 (75250.93)
  AUC0-24 | 41637.2 (24361.51) | 92527.5 (41122.30) | 171551.0 (75242.59)

23. Secondary Outcome: Pharmacokinetics of SB-497115-GR, CL/F
Description: CL/F: CL is an estimate of the total body clearance, and F is the fraction of dose absorbed.
Time Frame: Week 9 or 10
Population: PK Population. Data from one participant were abnormal; this participant was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: L/hr (Liters/hour)
Groups:
- SB-497115-GR 25 mg: Participants who received 25 mg of SB497511-GR on the PK sampling day
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 7 | 5 | 4
L/hr (Liters/hour) | 0.37156 (0.154284) | 0.30923 (0.114096) | 0.33035 (0.124401)

24. Secondary Outcome: Pharmacokinetics of SB-497115-GR, Vz/F
Description: VZ/F: VZ is the volume of distribution based on the terminal phase, and F is the fraction of dose absorbed.
Time Frame: Week 9 or 10
Population: PK Population. Data from one participant were abnormal; this participant was excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- SB-497115-GR 50 mg: Participants who received 50 mg of SB497511-GR on the PK sampling day
Arm/Group | SB-497115-GR 12.5 mg | SB-497115-GR 25 mg | SB-497115-GR 50 mg
Number analyzed (Participants) | 7 | 5 | 4
Liters | 5.6267 (2.00964) | 5.3870 (1.75077) | 5.0391 (1.76091)

ADVERSE EVENTS:
Time Frame: AE data were collected from the beginning of the double-blind (DB) phase. In the Long-Term (LT) phase, AEs were pooled from all participants (pts) who started the DB phase, regardless of whether they completed the phase.
Description: Participants (pts) taking placebo in the DB phase took SB-497115-GR (drug) in the OL phase for up to 26 weeks (wks). Pts receiving drug in the DB phase for 7 wks continued to receive it in the OL phase for 19 wks. Data from the 2 groups were pooled as a 26-wk treatment of drug for analysis. Thus, 23 pts were at risk in the Long-Term Phase.
Groups:
- Placebo Short-Term (Double-Blind) Phase: Placebo 12.5 mg for the first 3 weeks of the double-blind phase. The dose of placebo was adjusted at Week 3 based on the participant's platelet count and then continued up to Week 7.
- SB-497115-GR Short-Term (Double-Blind) Phase: SB-497115-GR 12.5 mg for the first 3 weeks of the double-blind phase. The dose of study medication was adjusted at Week 3 based on the participant's platelet count and then continued up to Week 7.
- SB-497115-GR Long-Term Phase: All participants who received placebo and SB-497115-GR in the double-blind phase and completed the phase continued to receive SB-497115-GR in the open-label phase (19 weeks for SB-497115-GR group and 26 weeks for placebo group; all participants received up to 26 weeks in total). Dose adjustment to 12.5, 25, or 50 mg/day was allowed based on the participant's platelet count
Arm/Group | Placebo Short-Term (Double-Blind) Phase | SB-497115-GR Short-Term (Double-Blind) Phase | SB-497115-GR Long-Term Phase
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/15 | 6/23
Other Adverse Events (participants affected / at risk) | 2/8 | 7/15 | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Short-Term (Double-Blind) Phase (N=8) | SB-497115-GR Short-Term (Double-Blind) Phase (N=15) | SB-497115-GR Long-Term Phase (N=23)
Hemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 2
Transient ischemic attack (Nervous system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Short-Term (Double-Blind) Phase (N=8) | SB-497115-GR Short-Term (Double-Blind) Phase (N=15) | SB-497115-GR Long-Term Phase (N=23)
Nasopharyngitis (Infections and infestations) | 0 | 4 | 10
Alanine aminotransferase increased (Hepatobiliary disorders) | 0 | 3 | 4
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 | 1 | 3
Headache (Nervous system disorders) | 1 | 1 | 3
Cystitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Herpes simplex (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Platelet count increased (Blood and lymphatic system disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 2
Conjunctival hemorrhage (Eye disorders) | 0 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Cataract (Eye disorders) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase decresed (Investigations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Cystitis-like symptom (Renal and urinary disorders) | 0 | 1 | 0
Dysmenorrhoea (Renal and urinary disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.